CLINICAL TRIAL: NCT01918189
Title: Development of an Internet-based Behavioral Pain Management Intervention
Brief Title: Internet-based Behavioral Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0998-R
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Chronic Low Back Pain
Keywords: back pain; low back pain; chronic pain; cognitive behavior therapy; behavior therapy
MeSH Terms: conditions — Back Pain; Low Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 10 week Pain EASE access (Experimental): behavioral pain self-management intervention (Pain EASE) delivered via the Internet
  Interventions: Behavioral: behavioral pain self-management intervention Pain EASE

INTERVENTIONS:
Behavioral: behavioral pain self-management intervention Pain EASE — 10 modules describing behavioral and cognitive pain coping skills such as relaxation and stress reduction methods, exercise and structured physical activity, and activity pacing

SUMMARY:
The purpose of the proposed project is to develop and test how well an internet-based behavioral pain self-management program, the Pain EASE program, can be used for treating low back pain in Veterans. Veterans' experiences with usability and satisfaction with the Pain EASE program will also be examined. Behavioral interventions such as exercise and cognitive behavior therapy are known to be effective for low back pain but are often not readily available or easily accessed. Veterans will be able to access the Pain EASE program via their computer with an internet connection, which will increase access to this type of treatment. Study participants will receive 10 weeks of access to the Pain EASE program, which will teach them pain coping skills to manage their low back pain. The primary outcome is pain-related functional interference.

DETAILED DESCRIPTION:
OBJECTIVES: The primary objectives of the proposed study are to: (1) develop an integrative, Internet-based, Veteran-centered behavioral intervention, the Pain EASE program for chronic low back pain (CLBP), and (2) examine preliminary efficacy, usability, and satisfaction of this intervention in a representative sample of Veterans with CLBP. The primary hypothesis states that a clinically meaningful reduction in pain-related functional interference will be observed following ten weeks of exposure to the Pain EASE program relative to baseline. The secondary hypotheses state that clinically meaningful reductions in ratings of average pain intensity on a 0 (no pain) to 10 (worst pain imaginable) numeric rating scale at the ten week post-baseline follow-up assessment interval will be observed, in addition to statistically significant reductions in fatigue, sleep problems, depressive symptoms, and negative mood at the ten week post-baseline assessment. The tertiary hypotheses state that participants will report high levels of interest, site usage, and satisfaction.

RESEARCH DESIGN: A non-randomized pilot study with two phases is proposed to develop and evaluate an internet-based behavioral pain self-management program. Phase I will solely involve qualitative data collection. Repeated quantitative assessments during Phase II will be conducted at baseline and 10-weeks post-baseline.

METHODOLOGY: A 24-month pilot study with two phases is proposed. During Phase I, the Pain EASE program will be developed and feedback from 15 Veterans with CLBP and an Expert Panel of pain management clinicians will be used to modify the program. During Phase II, a pilot feasibility trial of the Pain EASE program with 55 Veterans with CLBP will be conducted. Subjects will be a total of 70 patients receiving care at the VA Connecticut Healthcare System (VACHS) who report chronic low back pain. The primary criteria for inclusion are constant pain of at least three months duration with at least a moderate level of average pain (i.e., scores of 4 or greater on a 0 [no pain] to 10 [worst pain imaginable]) on a numerical rating scale of pain and indication of the "preparation", "action", or "maintenance" stage of readiness to change on a brief five item staging checklist. All patients must have access to a computer with an internet connection. Excluded will be patients with life threatening or acute physical illness, current alcohol or substance abuse or dependence, current psychosis, suicidal ideation, dementia, and individuals seeking surgical pain treatment. All participants will continue to receive their usual care from Veterans Health Administration (VHA) providers. During the 10-week therapeutic window, weekly telephone calls from research staff will serve to cue and monitor participants' use of the Internet program. At ten weeks post-baseline, participants will be formally reassessed. Primary and secondary hypotheses involving quantitative data will be analyzed using an intent-to-treat principle and will employ t-tests and non-parametric analogs and regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least a moderate level of chronic low back pain (i.e., numeric rating scale pain scores of 4) and presence of low back pain for a period of 3 months;
* Availability of a computer with Internet access;
* Indication of the "preparation", "action", or "maintenance" stage of readiness to change on a brief five item staging checklist and a rating of at least 4 or greater on a 0 (not at all interested) to 10 (extremely interested) rating scale designed to ensure participants' interest in receiving pain self-management via the Internet;
* Veteran receiving care at VA Connecticut Healthcare System

Exclusion Criteria:

* life threatening or acute medical condition that could impair participation (e.g., severe COPD, lower limb amputation, terminal cancer);
* psychiatric condition (e.g., active substance abuse, psychosis or suicidality) that could impair participation
* surgical interventions for pain during their participation in this study
* sensory deficits that would impair participation (e.g., visual impairment affecting ability to navigate Internet-based intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M. Higgins, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reuman L, Solar C, MacLean RR, Halat AM, Rajeevan H, Williams DA, Heapy AA, Bair MJ, Krein SL, Kerns RD, Higgins DM. If you personalize it, will they use it?: Self-reported and observed use of a tailored, internet-based pain self-management program. Transl Behav Med. 2022 May 26;12(5):693-701. doi: 10.1093/tbm/ibab165. PMID 35192703
- [Derived] Higgins DM, Buta E, Williams DA, Halat A, Bair MJ, Heapy AA, Krein SL, Rajeevan H, Rosen MI, Kerns RD. Internet-Based Pain Self-Management for Veterans: Feasibility and Preliminary Efficacy of the Pain EASE Program. Pain Pract. 2020 Apr;20(4):357-370. doi: 10.1111/papr.12861. Epub 2020 Jan 28. PMID 31778281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began July 1, 2014 and last data collection for primary outcome was October 31, 2018. Recruitment target of 58 participants was met. 59 participants enrolled in the study (i.e., signed informed consent) but 58 completed baseline measures and were included in outcomes analyses.
Period: Overall Study
Arm/Group | 10 Week Pain EASE Access
Started (59 participants enrolled (i.e., signed informed consent) but 58 completed baseline assessment.) | 59
Completed Baseline Assessment | 58
Completed Follow-up Assessment | 41
Completed | 41
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: 59 participants enrolled in the study (i.e., signed informed consent) but 58 completed baseline measures and were included in outcomes analyses.
Arm/Group | 10 Week Pain EASE Access
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 35
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58
Multidimensional Pain Inventory Interference Subscale [Mean (Standard Deviation); unit: units on a scale] — The 9-item Interference subscale, scores ranging from 0-6, of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI)-Interference scale assesses pain-related interference. A reduction in WHYMPI-Interference Scale scores of 0.6 or greater has been identified as an indicator of meaningful improvement in physical functioning.
  units on a scale | 3.82 (0.19)
Pain Intensity Numeric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — This is a likert scale self-report measures. Participants are asked, "Please rate your pain by indicating the number that best describes your average pain over the past week on a 0 (no pain) to 10 (pain as bad as you can imagine) scale". Scores of 1-3 reflect mild pain, 4-6 moderate pain, and 7-10 severe pain.
  units on a scale | 5.91 (0.25)
Profile of Mood States [Mean (Standard Deviation); unit: units on a scale] — Total mood symptoms score reported. The 65-item Profile of Mood States (POMS) is a multidimensional measure of emotional functioning designed to assess six dimensions of mood. Total Mood Disturbance score ranges from -32 to 200. Higher scores reflect poorer functioning.
  units on a scale | 49.53 (5.62)
Multidimensional Fatigue Inventory [Mean (Standard Deviation); unit: units on a scale] — Fatigue was assessed using the Multidimensional Fatigue Inventory (MFI), which is a 20 item measure that can be scored to produce 5 dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and how subscale statements regarding fatigue represent their experiences. Score range from 4 to 20. Higher total scores correspond with more acute levels of fatigue.
  units on a scale | 14.05 (0.52)
Medical Outcomes Study Sleep Scale [Mean (Standard Deviation); unit: units on a scale] — The MOS Sleep Scale is a 12 item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, awaken short of breath or with headache, adequacy of sleep, somnolence, a problems index 1 and a problems index 2). An additional single item assesses quantity of sleep. The sleep domains and problems index are scored on a 0-100 possible range, and higher scores indicate more of the concept being measured.
  units on a scale | 50.09 (3.80)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Depressive symptom severity was assessed using the 21-item Beck Depression Inventory. Scores range from 0 - 63. Higher scores indicate more severe depression symptomatology.
  units on a scale | 15.47 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Pain Inventory Interference Subscale
Description: Self-report measure of pain-related functional interference. The 9-item Interference subscale, scores ranging from 0-6, of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI)-Interference scale assesses pain-related interference. Lower scores indicate less pain-related interference (i.e., better outcome). A reduction in WHYMPI-Interference Scale scores of 0.6 or greater has been identified as an indicator of meaningful improvement in physical functioning.
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Population: 17 of the 58 participants who completed baseline did not complete 10-week post-baseline assessment (study endpoint)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 10 Week Pain EASE Access
Number analyzed (Participants) | 41
score on a scale | 0.53 [0.15 to 0.92]
Statistical Analysis 1: Comparison: 10 Week Pain EASE Access; Test type: Other — Mixed models (using an unstructured correlation structure) regression over the baseline and 10-week post-baseline follow-up assessments were used to examine change in outcome measures for preliminary efficacy variables. The primary endpoint for the preliminary efficacy analyses is the mean difference in baseline to post-baseline follow-up scores on the primary measure of pain interference (i.e., WHYMPI-Interference Scale) at 10 weeks post-baseline; p = 0.008, Regression, Logistic — a priori threshold for statistical significance is p <0.05

2. Secondary Outcome: Numeric Rating Scale of Pain Intensity
Description: self-report measure of pain intensity measured on a 0-10 likert scale. Participants are asked, "Please rate your pain by indicating the number that best describes your average pain over the past week on a 0 (no pain) to 10 (pain as bad as you can imagine) scale". Scores of 1-3 reflect mild pain, 4-6 moderate pain, and 7-10 severe pain. Lower scores reflect less pain, and therefore, better outcome.
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Behavioral Pain Self-management Intervention (Pain EASE): 10 weeks access to behavioral pain self-management intervention (Pain EASE) for low back pain delivered via the Internet
Arm/Group | Behavioral Pain Self-management Intervention (Pain EASE)
Number analyzed (Participants) | 41
units on a scale | -0.24 [-0.29 to 0.20]
Statistical Analysis 1: Comparison: Behavioral Pain Self-management Intervention (Pain EASE); Test type: Other — Mixed models (using an unstructured correlation structure) regression over the baseline and 10-week post-baseline follow-up assessments were used to examine change in outcome measures for preliminary efficacy variables. The primary endpoint for the preliminary efficacy analyses is the mean difference in baseline to post-baseline follow-up scores on the primary measure of pain intensity at 10 weeks post-baseline; p = 0.27, Regression, Logistic — a priori threshold for statistical significance is p<0.05; Mean Difference (Final Values) = 0.05

3. Secondary Outcome: Profile of Mood States
Description: Total mood symptoms score reported. The 65-item Profile of Mood States (POMS) is a multidimensional measure of emotional functioning designed to assess six dimensions of mood "over the past week, including today". Each item is scored on a 0-5 Likert scale, where 0= "not at all" and 5= "extremely". Total Mood Disturbance score ranges from 0 to 200. Higher scores reflect poorer functioning. Lower scores correspond to better outcomes.
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral Pain Self-management Intervention (Pain EASE)
Number analyzed (Participants) | 41
score on a scale | -9.57 [-17.72 to -1.42]
Statistical Analysis 1: Comparison: Behavioral Pain Self-management Intervention (Pain EASE); Test type: Other — Mixed models (using an unstructured correlation structure) regression over the baseline and 10-week post-baseline follow-up assessments were used to examine change in outcome measures for preliminary efficacy variables. The primary endpoint for the preliminary efficacy analyses is the mean difference in baseline to post-baseline follow-up scores on the measure of mood symptoms at 10 weeks post-baseline; p = 0.02, Regression, Logistic — a priori threshold for statistical significance is p<0.05; Mean Difference (Net) = 0.05

4. Secondary Outcome: Multidimensional Fatigue Inventory
Description: General fatigue scale reported. Fatigue was assessed using the Multidimensional Fatigue Inventory (MFI), which is a 20 item measure that can be scored to produce 5 dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and how subscale statements regarding fatigue represent their experiences. Score range from 4 to 20. Higher total scores correspond with more acute levels of fatigue. Lower scores correspond to better outcomes.
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral Pain Self-management Intervention (Pain EASE)
Number analyzed (Participants) | 41
score on a scale | -0.3 [-1.17 to 0.56]
Statistical Analysis 1: Comparison: Behavioral Pain Self-management Intervention (Pain EASE); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.48, Regression, Logistic — a priori threshold for statistical significance is p<0.05; Mean Difference (Net) = 0.05

5. Secondary Outcome: Medical Outcomes Study Sleep Scale
Description: The MOS Sleep Scale is a 12 item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, awaken short of breath or with headache, adequacy of sleep, somnolence, a problems index 1 and a problems index 2). An additional single item assesses quantity of sleep. The sleep domains and problems index are scored on a 0 - 100 possible range, and higher scores indicate more of the concept being measured. Lower scores on sleep disturbance, for example, reflect less disturbed sleep, which is a better outcome.
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral Pain Self-management Intervention (Pain EASE)
Number analyzed (Participants) | 41
score on a scale | -4.95 [-12.27 to 2.38]
Statistical Analysis 1: Comparison: Behavioral Pain Self-management Intervention (Pain EASE); Test type: Other — Mixed models (using an unstructured correlation structure) regression over the baseline and 10-week post-baseline follow-up assessments were used to examine change in outcome measures for preliminary efficacy variables. The primary endpoint for the preliminary efficacy analyses is the mean difference in baseline to post-baseline follow-up scores on the measure of sleep at 10 weeks post-baseline; p = 0.18, Regression, Logistic — a priori threshold for statistical significance is p<0.05; Mean Difference (Net) = 0.05

6. Secondary Outcome: Beck Depression Inventory
Description: Depressive symptom severity was assessed using the 21-item Beck Depression Inventory. Scores range from 0 - 63. Higher scores indicate more severe depression symptomatology. Lower scores correspond to better outcomes (i.e., less depressive symptom severity).
  Outcome was calculated as a change from baseline score to 10-week post-baseline score (i.e., 10 weeks post-baseline value minus baseline value).
Time Frame: baseline and 10 weeks post-baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral Pain Self-management Intervention (Pain EASE)
Number analyzed (Participants) | 41
score on a scale | -2.31 [-4.37 to -0.25]
Statistical Analysis 1: Comparison: Behavioral Pain Self-management Intervention (Pain EASE); Test type: Other — Mixed models (using an unstructured correlation structure) regression over the baseline and 10-week post-baseline follow-up assessments were used to examine change in outcome measures for preliminary efficacy variables. The primary endpoint for the preliminary efficacy analyses is the mean difference in baseline to post-baseline follow-up scores on the measure of depression symptoms at 10 weeks post-baseline; p = 0.03, Regression, Logistic — a priori threshold for statistical significance is p<0.05; Mean Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: 10 weeks of active study participation
Groups:
- 10 Week Pain EASE Access: behavioral pain self-management intervention (Pain EASE) for chronic low back pain delivered via the Internet
  behavioral pain self-management intervention Pain EASE: 10 modules describing behavioral and cognitive pain coping skills such as relaxation and stress reduction methods, exercise and structured physical activity, and activity pacing
  Access to the Pain EASE intervention for 10 weeks: analyses were conducted to determine change from baseline on pain-related functional interference and other outcomes
Arm/Group | 10 Week Pain EASE Access
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 1/58
Other Adverse Events (participants affected / at risk) | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Week Pain EASE Access (N=58)
psychiatric emergency room visit (Psychiatric disorders) | 1 (1) — psychiatric emergency room visit for manic episode in the context of bipolar disorder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT01918189/Prot_SAP_000.pdf